CLINICAL TRIAL: NCT06882070
Title: ROTA-biotic: Measuring the Impact of Rotavirus Vaccines on Paediatric Antibiotic Usage
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Wellcome Trust (Other); Centre for Infectious Disease Research in Zambia (Other); Noguchi Memorial Institute for Medical Research (Other); Amsterdam Institute for Global Health and Development (Other)
Responsible Party: Principal Investigator, Vanessa Harris, Doctor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 219775/Z/19/Z
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-12

CONDITIONS: Rotavirus Gastroenteritis; Rotavirus Vaccines; Antimicrobial Resistance (AMR); Antibiotic; Microbiome; Infant Diarrhea
MeSH Terms: conditions — Diarrhea, Infantile | interventions — Vaccines; Vaccines, Attenuated; RIX4414 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Stool and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Trial cohort: This group received either the trivalent P2-VP8 subunit rotavirus vaccine or oral live attenuated vaccine, Rotarix®,
  Interventions: Other: Vaccine
- Community cohort: This acted as control group, away from the vaccine trial groups

INTERVENTIONS:
Other: Vaccine — Trivalent P2-VP8 subunit rotavirus vaccine
  Other Names: trivalent P2-VP8 subunit rotavirus vaccine; oral live attenuated vaccine, Rotarix®
  Groups: Trial cohort

SUMMARY:
Rotavirus is the most common aetiology of serious diarrhoea in young children. Despite antibiotics not being indicated in its treatment, diarrhoea remains a very common cause for antibiotic prescribing in low-income settings. We hypothesized that effective rotavirus vaccination could reduce diarrhoeal episodes and thereby unnecessary antibiotic usage in young children in low-income settings.

The study aimed to evaluate the impact of rotavirus vaccination on antibiotic usage. Specifically, the study quantified how differences in rotavirus vaccine efficacy would impact days of prescription and nonprescription antibiotic usage in the first 2 years of life among two large cohorts of children in Zambia and Ghana.

The key goal was to understand the effect of rotavirus vaccine efficacy on antibiotic usage and household antibiotic costs. The goal was to generate evidence needed to inform policymakers seeking to introduce new rotavirus vaccines into national vaccination programs, of potential, and often under-appreciated, secondary effects of rotavirus vaccine implementation on antibiotic usage.

The study was conducted within a Phase III randomised controlled trial comparing the efficacy of a new parenteral trivalent P2-VP8 subunit rotavirus vaccine to the oral live attenuated vaccine, Rotarix®, against severe rotavirus gastroenteritis in the first 2 years of life in Zambia and Ghana.

ELIGIBILITY:
Inclusion Criteria:

Healthy infants as established by medical history and clinical examination before randomisation into the study Age: ≥6 and <8 weeks at the time of first study vaccination (42 days through 55 days old, inclusive, with the day after birth considered 1-day old) Parental ability and willingness to provide written informed consent. Intention of the participants' parents to remain in the area with the child during the study period

Exclusion Criteria:

Acute disease at the time of enrollment/first study vaccination - temporary exclusion Presence of fever on the day of enrollment/first study vaccination (axillary temperature >37.6oC) Concurrent participation in another clinical trial (other than the parent study) throughout the entire timeframe for this study.

Presence of severe malnutrition (weight-for-height z-score ≤-3SD median (per WHO published child growth standards) History of premature birth (<37 weeks gestation) and/or birth weight of <2.5 kg History of congenital abdominal disorders, intussusception, or abdominal surgery Prior receipt of rotavirus vaccine

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The infants were from communities that are typical peri-urban settlements in Zambia and Ghana with informal housing, poor sanitation and mostly shared water supply from communal boreholes. These were high density communities with high unemployment rates and generally high incidence of infectious diseases.
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
To assess the relative efficacy of the TV P2-VP8 vaccine in comparison to Rotarix® in reducing prescription and non-prescription antibiotic consumption in the first two years of life. | 2 years

SECONDARY OUTCOMES:
• To assess the relative efficacy of the TV P2-VP8 vaccine in comparison to Rotarix® in reducing recurrent antibiotic consumption in the first two years of life. | 2 years
• To assess the relative efficacy of the TV P2-VP8 vaccine in comparison to Rotarix® in reducing household prescription and non-prescription antibiotic costs in the first two years of life. | 2 years
• To assess the background incidence of antibiotic usage in the community in the first two years of life. | 2 years
• To assess the relationship between frequency of antibiotic use and faecal bacterial microbiome composition, ARG abundance and bacterial metabolites in the urine over the first two years of life. | 2 years
• To assess the relationship between RVV efficacy (TV P2-VP8 and Rotarix) and faecal bacterial microbiome composition over the first two years of life. | 2 years
• Verification of weekly recall and medicine cabinet review of antibiotic use through assessment of antibiotic metabolites in the urine. | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Noguchi Memorial Institute of Medical Research-University of Ghana, Accra, Ghana
- Center for Infectious Disease Research in Zambia, Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: Undecided